CLINICAL TRIAL: NCT03519243
Title: Randomized Open-Label Comparative Study of the Efficacy and Safety of BCD-131 (JSC BIOCAD, Russia) and Mircera (F. Hoffmann-La Roche Ltd, Switzerland) in Treatment of Anemia in Chronic Kidney Disease Patients on Dialysis
Brief Title: Comparative Study of the Efficacy and Safety of BCD-131 and Mircera in Treatment of Anemia in CKD Patients on Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCD-131-2
Record Dates: First submitted 2018-04-26; First posted 2018-05-08 (Actual); Results first posted 2019-07-26 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BCD-131 1,05 mcg/kg * conversion ratio (Experimental): subcutaneously monthly
  Interventions: Biological: BCD-131
- BCD-131 1,7 mcg/kg * conversion ratio (Experimental): subcutaneously monthly
  Interventions: Biological: BCD-131
- BCD-131 2,75 mcg/kg * conversion ratio (Experimental): Subcutaneously monthly
  Interventions: Biological: BCD-131
- Mircera (Active Comparator): subcutaneously monthly
  Interventions: Biological: Mircera

INTERVENTIONS:
Biological: BCD-131 — subcutaneously monthly
  Other Names: pegylated darbepoetin beta
  Arms: BCD-131 1,05 mcg/kg * conversion ratio; BCD-131 1,7 mcg/kg * conversion ratio; BCD-131 2,75 mcg/kg * conversion ratio
Biological: Mircera — subcutaneously monthly
  Other Names: Methoxy polyethylene glycol-epoetin beta
  Arms: Mircera

SUMMARY:
BCD-131 is pegylated darbepoetin beta. BCD-131-2 is International Multicenter Randomized Open-Label Comparative Study (Phase II) of the Efficacy and Safety of BCD-131 and Mircera in Treatment of Anemia in Chronic Kidney Disease Patients on Dialysis.

DETAILED DESCRIPTION:
The hypothesis of the study is that the efficacy of BCD-131 is equivalent to that of Mircera® based on the analysis of the primary endpoint (changes in the Hb level over the period of evaluation as compared to the baseline Hb level ) during the 21-week period of treatment.

This study is a study of the maintenance treatment of anemia. The study will include up to 100 dialysis patients with stage 5D chronic kidney disease, established efficacy of dialysis and renal anemia without other causes of anemia, receiving erythropoiesis-stimulating agents (ESA) and reaching target hemoglobin levels.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Men and women aged from 18 to 75 years (inclusive) on the day of signing informed consent;
* End-stage kidney disease.
* Need for dialysis for at least 3 months before signing informed consent.
* Need for at least 12 hours on standard dialysis procedure weekly.
* rHuEpo (epoetin alpha, epoetin beta, darbepoetin alpha) administration for at least 3 months before signing informed consent.
* Regular rHuEpo (epoetin alfa, epoetin beta, darbepoetin alfa) administration 1, 2 or 3 times a week (stable dose, stable frequency) before signing informed consent.
* Target hemoglobin level (100-120 g/l) for at least 3 months before signing informed consent.
* Effective dialysis dose index (Kt/v) ≥1.2 for patients receiving hemodialysis and (Kt/v) ≥1.7 for patients receiving peritoneal dialysis.
* TSAT ≥20%, Serum ferritin >200 ng/ml.
* Patients and their sexual partners with childbearing potential must implement reliable contraceptive measures during all the study treatment, starting 4 weeks prior to the administration of the first dose of investigational product until 4 weeks after the last dose of investigational product. This requirement does not apply to participants who have undergone surgical sterilization. Reliable contraceptive measures include two methods of contraception, including one barrier method/
* Patients should be able to follow the Protocol procedures

Exclusion Criteria:

* Any other causes of anemia except for renal anemia, including folate and B12 deficiency, chronic blood loss, aluminium intoxication, sickle-cell anemia, chronic disease anemia (CRP above 20 mg/l), refractory anemia with blast cells in peripheral blood.
* Lupus nephritis of kidney disease due to systemic vasculitis.
* Platelet count below 100х10^9 cells/l.
* Scheduled kidney transplant during study participation period.
* Hypersensitivity to darbepoetin alfa or of any components of study drugs, or to Fe (III)-hydroxide-sucrose complex.
* Vaccination less than 8 weeks before signing informed consent.
* Liver cirrhosis with portal hypertension and/or splenomegaly and/or ascitis.
* HIV infection, active HBV, HCV.
* ALT, AST level above 3x ULN.
* Congestive heart failure (Grade IV NYHA)
* Resistant arterial hypertension.
* Unstable angina.
* Hemoglobinopathy, MDS, hematologic malignancy, PRCA.
* Severe secondary hyperparathyroidism.
* Gastrointestinal bleeding history.
* Thrombotic events history (myocardial infarction, stroke, TIA, DVT, PATE) less than 6 months before signing informed consent.
* Seizures, including epilepsy.
* Major surgery in less than 1 month before signing informed consent
* Blood transfusions in less than 3 months before signing informed consent.
* Acute inflammatory diseases or exacerbations of chronic inflammation.
* Severe psychiatric disorders and suicidal ideation and suicidal behavior.
* History of malignancy, excluding appropriately treated basal cell carcinoma or cervical carcinoma in situ.
* Alcohol or drug abuse.
* Simultaneous participation in other trials or in less than 3 months before signing informed consent
* Pregnancy of breast-feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JCS BIOCAD
Locations (3):
- City Clinical Hospital №9, Minsk, Belarus
- Russia (2):
  - City Mariin Hospital, Saint Petersburg
  - B.Braun Avitum Russland Clinics Ltd., Saint Petersburg

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BCD-131 1,05 mcg/kg * Conversion Ratio | BCD-131 1,7 mcg/kg * Conversion Ratio | BCD-131 2,75 mcg/kg * Conversion Ratio | Mircera
Started | 25 | 25 | 0 (The dose level was not studied due to the dose level l.7 µg/kg demonstrated the sufficient PD effect) | 25
Completed | 20 | 21 | 0 | 24
Not Completed | 5 | 4 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BCD-131 1,05 mcg/kg * Conversion Ratio | BCD-131 1,7 mcg/kg * Conversion Ratio | Mircera | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [48 to 64] | 54 [46 to 63] | 47 [35 to 58] | 55 [46 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 11 | 37
  Male | 11 | 13 | 14 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 24 | 25 | 24 | 73
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Belarus | 5 | 1 | 2 | 8
  Russia | 20 | 24 | 23 | 67

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin (Hb) Concentration From Baseline to the Evaluation Period
Description: The baseline hemoglobin will be calculated as the arithmetic mean of hemoglobin values obtained at screening and at Visit 1. The final hemoglobin value during the evaluation period will be calculated as the arithmetic mean of hemoglobin values obtained at Week 21 and Week 23.
Time Frame: Baseline - measurements on Screening (weeks -4 - 0) and on day 1; Evaluation period - weekly measures on weeks 21 to 23
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | BCD-131 1,05 mcg/kg * Conversion Ratio | BCD-131 1,7 mcg/kg * Conversion Ratio | Mircera
Number analyzed (Participants) | 20 | 21 | 24
g/L | -3.25 [-12 to 0.5] | 3.5 [-7 to 14] | -2.75 [-9.5 to 9]

2. Secondary Outcome: The Proportion of Patients Who Developed AEs/SAEs That, in the Investigator's Opinion, Are Related to BCD-131
Description: The proportion of patients, in each group, who developed СТСАЕ v. 4.03 Grade 3-4 AEs that, in the Investigator's opinion, are related to BCD-131
  - the proportion of patients, in each group, who discontinued the study due to AEs/SAEs
Time Frame: Week 23
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-131 1,05 mcg/kg * Conversion Ratio | BCD-131 1,7 mcg/kg * Conversion Ratio | Mircera
Number analyzed (Participants) | 25 | 25 | 25
Participants | 5 | 2 | 2

3. Secondary Outcome: The Proportion of BAb- and NAb-positive Patients
Description: Blood sampling for immunogenicity assessment (BAbs and NAbs) will be performed in all the patients included in the study before the first injection and then at Week 9 and Week 23.
  The immunogenicity endpoints will be analyzed after the completion of all periods of the study.
Time Frame: Week 9, 23
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-131 1,05 mcg/kg * Conversion Ratio | BCD-131 1,7 mcg/kg * Conversion Ratio | Mircera
Number analyzed (Participants) | 24 | 25 | 25
Participants | 0 | 0 | 0

4. Secondary Outcome: AUC(0-672 Hour)
Description: Area under the concentration curve from the moment of injection to 672 h [28 days])
Time Frame: 3, 6, 12, 24, 48, 72, 96, 168, 336, 504, 672 h h after injection 1
Measure: Median (Inter-Quartile Range); unit: (mmol/L)*h
Arm/Group | BCD-131 1,05 mcg/kg * Conversion Ratio | BCD-131 1,7 mcg/kg * Conversion Ratio | Mircera
Number analyzed (Participants) | 15 | 15 | 15
(mmol/L)*h | 51744.45 [31201.8 to 87463.5] | 73948.8 [57057.15 to 133730.25] | 89409.3 [35389.95 to 166699.5]

5. Secondary Outcome: AUC(0-∞)
Description: Area under the concentration curve from the moment of injection to infinity
Time Frame: 3, 6, 12, 24, 48, 72, 96, 168, 336, 504, 672 h h after injection 1, weeks 5, 9, 13, 17, 21
Measure: Median (Inter-Quartile Range); unit: (mmol/L)*h
Arm/Group | BCD-131 1,05 mcg/kg * Conversion Ratio | BCD-131 1,7 mcg/kg * Conversion Ratio | Mircera
Number analyzed (Participants) | 15 | 15 | 15
(mmol/L)*h | 65150.045 [43463.791 to 91305.66] | 81698.001 [63442.206 to 142665.693] | 96259.513 [46985.695 to 192570.672]

6. Secondary Outcome: Cmax
Description: Maximum serum concentration of the drug product) after the first injection of the test/reference drug
Time Frame: 3, 6, 12, 24, 48, 72, 96, 168, 336, 504, 672 h h after injection 1, weeks 5, 9, 13, 17, 21
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | BCD-131 1,05 mcg/kg * Conversion Ratio | BCD-131 1,7 mcg/kg * Conversion Ratio | Mircera
Number analyzed (Participants) | 15 | 15 | 15
mmol/L | 195.3 [148.7 to 407.1] | 231.9 [187.2 to 488.2] | 617.6 [130.6 to 943.2]

7. Secondary Outcome: AUEC(0-672 Hour)
Description: Area under the effect curve from the drug injection to 672 h [28 days]) based on the change in the absolute reticulocyte count after the first injection of the test/reference drug
Time Frame: 3, 6, 12, 24, 48, 72, 96, 168, 336, 504, 672 h h after injection 1
Measure: Mean (Standard Deviation); unit: (cells*10^9)*h
Arm/Group | BCD-131 1,05 mcg/kg * Conversion Ratio | BCD-131 1,7 mcg/kg * Conversion Ratio | Mircera
Number analyzed (Participants) | 15 | 15 | 15
(cells*10^9)*h | 7210.479 (5465.155) | 11274.380 (12460.177) | 12131.820 (15613.087)

8. Secondary Outcome: AC-Emax
Description: Maximum absolute reticulocyte count after the first injection of BCD-131/Mircera®
Time Frame: day 28
Measure: Mean (Standard Deviation); unit: (cells*10^9)/L
Arm/Group | BCD-131 1,05 mcg/kg * Conversion Ratio | BCD-131 1,7 mcg/kg * Conversion Ratio | Mircera
Number analyzed (Participants) | 15 | 15 | 15
(cells*10^9)/L | 96.650 (29.185) | 107.047 (38.615) | 154.753 (58.729)

ADVERSE EVENTS:
Time Frame: 25 weeks
Arm/Group | BCD-131 1,05 mcg/kg * Conversion Ratio | BCD-131 1,7 mcg/kg * Conversion Ratio | Mircera
All-Cause Mortality (participants affected / at risk) | 1/25 | 2/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 6/25 | 4/25 | 3/25
Other Adverse Events (participants affected / at risk) | 13/25 | 16/25 | 15/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCD-131 1,05 mcg/kg * Conversion Ratio (N=25) | BCD-131 1,7 mcg/kg * Conversion Ratio (N=25) | Mircera (N=25)
subcutaneous tissue (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Infection of postsurgical subcutaneous seroma
consequence of stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
fracture of the left ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischemic Heart Disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
non-Q wave myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous Access Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes. Diabetic foot syndrome (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter-associated infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Phlebitis of the fistula vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
arteriovenous fistula stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
acute gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCD-131 1,05 mcg/kg * Conversion Ratio (N=25) | BCD-131 1,7 mcg/kg * Conversion Ratio (N=25) | Mircera (N=25)
arterial pressure increase (Vascular disorders) | 4 (4) | 3 (3) | 3 (3)
lymphocytes decrease (Investigations) | 4 (4) | 2 (2) | 1 (1)
hyperglycemia (Investigations) | 6 (6) | 4 (4) | 2 (2)
leukocytes decrease (Investigations) | 2 (2) | 1 (1) | 1 (1)
neutrophils decrease (Investigations) | 2 (2) | 2 (2) | 2 (2)
ECG changes (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
lymphocytes increase (Investigations) | 1 (1) | 0 (0) | 2 (2)
systolic blood pressure increase (isolated) (Vascular disorders) | 3 (3) | 6 (6) | 4 (4)
dyastolic blood pressure increase (isolated) (Vascular disorders) | 2 (2) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT03519243/Prot_SAP_003.pdf